CLINICAL TRIAL: NCT02923908
Title: A Pilot Study of Facial Recognition Software to Assess Palatability in Pediatric Patients
Brief Title: Recording Facial Expressions to Assess Taste in Children and Teenagers
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: GK003; 20162192 (Other: Western Institutional Review Board)
Record Dates: First submitted 2016-09-30; First posted 2016-10-05 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Facial Expression
Keywords: Palatability; Pediatrics; Facial Recognition; Taste; Facial Expressions
MeSH Terms: conditions — Facial Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Using a sample of saliva or swabbed buccal mucosa, a given DNA sample will be analyzed for allelic variants of a gene (TAS2R38), which controls the expression of the bitter taste receptor in each subject. This analysis will be exploratory in nature and its value would be to investigate any potential genotype-phenotype discordance in a given participant in response to the bitter (Prednisone) test substance. The DNA samples will only be used to assess genomic interactions in taste response.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Noldus Facereader 7 — A video recording of a subject's facial expressions while tasting a sweet, bitter, and neutral flavored liquid will be analyzed using Noldus Facereader 7 software.
Other: Voice Recording — A voice recording will be made for the duration of the tasting period.
Other: 5-Point Facial Hedonic Scale — A 5-point facial hedonic scale will be given to the participant to complete prior to the administration of any test substances and about 5, 10, and 30 minutes after the administration of each test substance.
Other: Follow-Up Questionnaire — Participants will be asked a few questions about each test agent after tastings.

SUMMARY:
The study is designed to see if, after tasting specific things, whether a child's facial pattern and voice pattern can determine the difference in something that has a sweet taste, no taste, and a bitter taste. The investigators will do this by comparing video recordings of a child's facial expression and voice to the child's response to follow-up questions after tasting three (3) different substances.

DETAILED DESCRIPTION:
Participants will taste three different substances in random order: 1. Prednisone liquid (a commonly used medicine to treat swelling which is approved by the Food and Drug Administration) for use in children; 2. A solution of table sugar in water (simple syrup); and 3. Ora-Plus, which is a solution that can be added to medicines. Ora-Plus is considered safe for use in children's formulas and all of the ingredients of Ora-Plus are on the Food and Drug Administration (FDA) Generally Regarded as Safe (GRAS) list. About 1 ml of each substance will be placed directly onto the tongue. Each substance will be tasted for 5-10 seconds and then, expectorated. Participants and investigators recording responses will be blinded with regard to the identity of test substances.

Facial expression will be recorded prior to administration of the taste substances and for approximately 2 minutes thereafter. An audio recording of the participant's voice will also be made during this time. At about 5 and 10 minutes after a given taste substance is administered, participants will be asked to identify a face on a 5-point facial hedonic scale which shows the participant's taste perception. Participants will also be asked to describe the taste sensation experienced as sweet, bitter or neutral (no apparent taste).

Participants will have a 30-minute rest period after administration of each taste substance which will include the administration of water and a neutral food to enable cleansing of the palate. The procedure above will be repeated in the same way for each of the 3 test substances.

ELIGIBILITY:
Inclusion Criteria:

Participants will be eligible if all of the following criteria is met:

* Verbal assent and parental consent provided.
* Males and females between 7 and ≤16 years of age (n= 3-5 in group 7 to 11 years and n= 4-5 in group 12 to ≤16 years. An additional 3 participants may be recruited if a recording does not produce viable data.)
* Both parent and participant speak English proficiently

Exclusion Criteria:

Participants will not be eligible if any of the following criteria is met:

* Unwillingness to participate.
* Participants of Asian ethnicity (N.B. The current FaceReader software cannot correctly identify facial expressions in these children and as a result cannot produce an analysis suitable to this study.14)
* Any medical condition or recent event that would cause a study participant to be unable to taste or swallow study agents.
* Any medical condition, previous surgery, or recent event affecting the tongue or palate that would cause taste alteration or aversion (i.e. ulcerations or infection of the tongue, soft or hard palate).
* Any medical condition or recent event that would preclude a study participant from having an intact sense of smell (i.e. anosmia, history of severe sinus infections, recent upper respiratory infection with congestion).
* Had a dentist visit within 14 days prior to enrollment or the time between enrollment and receipt of study articles.
* Any history of allergy, hypersensitivity, or intolerance to prednisone, sugar, food dyes, or any of the constituents of Ora-Plus.
* Any prior history of cardiac or gastrointestinal problems with the exception of self-limited conditions common to pediatric patients.
* Have ingested any medication or food substance 60 minutes prior to administration of the test articles.
* If the participant is the child or a first-degree relative to any of the investigators.
* Any profound sensory deficit (i.e. vision or hearing) that may interfere with the ability to comply with study related demands.
* Neurocognitive Disorders that could limit interpretation of results and their generalizability.
* History of a chronic illness.
* Use of mouthwash within 24 hours of study visit.
* Participant does not pass the baseline medical assessment.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study participants will be recruited via IRB approved advertisements and from the ACRI database for which subjects have given prior permission to be contacted for research studies. A convenience sample will be comprised of 10 children and/or adolescents ranging in age from 7 to 16 years of age. A total of 13 subjects may be enrolled in the event that a subject is unable to meet criteria and/or needs to withdraw. If the study attains 10 evaluable subjects, then additional participants will not be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-12; Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Evidence that recording of facial expressions can reliably distinguish between liquids that taste bitter, sweet, or have no taste | within one year of study procedure
  The investigators propose that Noldus Facereader 7 can adequately discriminate between bitter, sweet, and neutral tastes in children and adolescents. Data collected through these recordings will be compared to ratings of liking/disliking of liquids using a 5-point facial hedonic scale and compared to a questionnaire after each tasting.

OTHER OUTCOMES:
Audio Recording During Study Procedure | within one year of study procedure
  An audio recording will occur during the tasting of each liquid in order to capture the subject's response to the liquid. This recording will be analyzed to determine a subject's liking/disliking of each test agent.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory L Kearns, PharmD, PhD, Principal Investigator — Arkansas Children's Research Institute
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available. However, the overall results of the study will be made available.

REFERENCES:
- [Background] Walsh J, Cram A, Woertz K, Breitkreutz J, Winzenburg G, Turner R, Tuleu C; European Formulation Initiative. Playing hide and seek with poorly tasting paediatric medicines: do not forget the excipients. Adv Drug Deliv Rev. 2014 Jun;73:14-33. doi: 10.1016/j.addr.2014.02.012. Epub 2014 Mar 12. PMID 24614069
- [Background] Matsui D. Current issues in pediatric medication adherence. Paediatr Drugs. 2007;9(5):283-8. doi: 10.2165/00148581-200709050-00001. PMID 17927300
- [Background] Wollner A, Lecuyer A, De La Rocque F, Sedletzki G, Derkx V, Boucherat M, Elbez A, Gelbert-Baudino N, Levy C, Corrard F, Cohen R. [Acceptability, compliance and schedule of administration of oral antibiotics in outpatient children]. Arch Pediatr. 2011 May;18(5):611-6. doi: 10.1016/j.arcped.2011.02.010. Epub 2011 Mar 21. French. PMID 21420838
- [Background] Winnick S, Lucas DO, Hartman AL, Toll D. How do you improve compliance? Pediatrics. 2005 Jun;115(6):e718-24. doi: 10.1542/peds.2004-1133. PMID 15930200
- [Background] Sjovall J, Fogh A, Huitfeldt B, Karlsson G, Nylen O. Methods for evaluating the taste of paediatric formulations in children: a comparison between the facial hedonic method and the patients' own spontaneous verbal judgement. Eur J Pediatr. 1984 Feb;141(4):243-7. doi: 10.1007/BF00572770. PMID 6734676
- [Background] Tolia V, Johnston G, Stolle J, Lee C. Flavor and taste of lansoprazole strawberry-flavored delayed-release oral suspension preferred over ranitidine peppermint-flavored oral syrup: in children aged between 5-11 years. Paediatr Drugs. 2004;6(2):127-31. doi: 10.2165/00148581-200406020-00006. PMID 15035653
- [Background] Mennella JA, Spector AC, Reed DR, Coldwell SE. The bad taste of medicines: overview of basic research on bitter taste. Clin Ther. 2013 Aug;35(8):1225-46. doi: 10.1016/j.clinthera.2013.06.007. Epub 2013 Jul 22. PMID 23886820
- [Background] Mennella JA, Reed DR, Roberts KM, Mathew PS, Mansfield CJ. Age-related differences in bitter taste and efficacy of bitter blockers. PLoS One. 2014 Jul 22;9(7):e103107. doi: 10.1371/journal.pone.0103107. eCollection 2014. PMID 25050705
- [Background] Danner, Lukas, Liudmila Sidorkina, Max Joechl, Klaus Duerrschmid. Make a face! Implicit and explicit measurement of facial expressions elicited by orange juices using face reading technology. Elsevier: Food Quality and Preference. 2013; 32:167-172.
- [Background] Loijens, Leanne, et. al. FaceReader: Reference Manual Version 7. Noldus Information Technology. Wageningen, 2016, pp. 55.
- See also: FDA Approval of Prednisone Oral Solution 5mg/5mL — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.DrugDetails